CLINICAL TRIAL: NCT03063697
Title: Prospective, Multi-center, Observational Study to Evaluate the Safety of DILATREND SR Cap. in Korean Patients With Essential Hypertension, Chronic Stable Angina and Congestive Heart Failure
Brief Title: Observational Study to Evaluate the Safety of DILATREND SR Cap. in Korean Patients With Essential Hypertension, Chronic Stable Angina and Congestive Heart Failure
Acronym: DELIGHT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 425HT15021
Record Dates: First submitted 2016-05-23; First posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Essential Hypertension; Chronic Stable Angina; Congestive Heart Failure
Keywords: Carvedilol SR Cap; Essential hypertension; Chronic stable angina; Congestive heart failure
MeSH Terms: conditions — Essential Hypertension; Angina, Stable; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients who check the safety data after taking Dilatrend SR

SUMMARY:
The purpose of this study is to Evaluate the Safety of DILATREND SR Cap. in Korean Patients with Essential hypertension, Chronic stable angina and Congestive heart failure for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 years or older Patients with Essential hypertension, Chronic stable angina and Congestive heart failure
2. Possible to take Dilatrend SR on the label
3. not taking Caverdilol for 6 month from Agreement date
4. Agreement with written informed consent

Exclusion Criteria:

1. Pregnancy or lactation
2. Known hypersensitivity to Carvedilol
3. Cardiogenic shock
4. Abnormality of the conduction system as Severe bradycardia(In particular, pulse <50beats / min), 2nd degree AV block, Complete AV block, Sinus Block, Sick Sinus Syndrome
5. Cor pulmonale
6. IDDM with ketoacidosis, metabolic acidosis
7. has severe heart disease(Heart failure NYHA functional class 4)
8. Respiratory diseases as Asthma, Chronic Obstructive Pulmonary Disease
9. Secondary hypertension
10. Prinzmetal's angina
11. Acute pulmonary embolism
12. Pheochromocytoma
13. Take MAO lnhibitor(except for MAO-B)
14. Hypotension ( SBP 90mmHg or less)
15. Severe hepatic dysfunction
16. Peripheral circulatory disturbance( ex. Raynaud syndrome, intermittent claudication)
17. Has edema glottitis
18. Has heart attack with complication
19. Fluid retention or overload to required intravenous inotropes
20. Allergic rhinitis

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: in Korean 20,000 Patients with Essential hypertension, Chronic stable angina and Congestive heart failure
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2015-11; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events and adverse drug reactions at 24 weeks | for 24 weeks
The incidence and severity of unexpected adverse events and adverse drug reactions at 24 weeks | for 24 weeks

IPD SHARING:
Plan to Share IPD: No